CLINICAL TRIAL: NCT05528497
Title: Assessment of the Influence of the Virtual Reality Headset on Pain and Anxiety During Oocyte Retrieval Under Local Anesthesia (OVOREV)
Brief Title: Assessment of the Influence of the Virtual Reality Headset on Pain and Anxiety During Oocyte Retrieval Under Local Anesthesia
Acronym: OVOREV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC22_8923_OVOREV; 2022-A01275-38 (Other: ANSM (N°ID-RCB))
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Oocyte Retrieval; Local Anaesthesia; Virtual Reality
Keywords: Oocyte Retrieval; Local anaesthesia; Virtual reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR+ (Experimental): For patients in the experimental group, using the virtual reality headset, the caregiver will place the headset on the patient as she is laid on the surgical table. The caregiver will ensure that the patient can see and hear the sequence that is being performed. The caregiver can then proceed to the different stages of ovocyte retrieval. Once the procedure is finished, the caregiver tells the patient that she can remove the headset
  Interventions: Other: VR+
- Control (No Intervention): For patients in the control group, without a headset, the oocyte retrieval procedure will not be modified.

INTERVENTIONS:
Other: VR+ — Use of a virtual reality helmet during ovocyte retrieval
  Arms: VR+

SUMMARY:
Medically Assisted Reproduction provides help to infertile couples, single women and couples of women with a pregnancy project, and to women who wish to preserve their gametes. In the context of In Vitro Fertilization (IVF), oocyte donation or oocyte preservation, it is necessary to perform an oocyte stimulation, followed by an ovarian puncture in order to retrieve mature oocytes. Several types of anesthesia can be used for this procedure: general anesthesia, local anesthesia and spinal anesthesia. The puncture can also be performed under hypnosis, but this practice is difficult to generalize, as it requires specific training. None of these different types of anesthesia has proven to be superior in terms of number and quality of oocytes collected, so the choice is left to the patient. General anesthesia is mostly chosen at Rennes, although it exposes to more risks and represents a higher socio-economic cost.

Improving the comfort of these patients during oocyte retrieval is a priority, especially since they may have to undergo several successive retrievals during their treatment. What if virtual reality could be a way to improve the comfort of these patients? Indeed, this technology, which allows activity in an artificial 3-dimensional world, is considered as a non-pharmacological tool for pain management and its use during surgery would also reduce the level of anxiety. In our study, during the oocyte retrieval under local anesthesia, the patients randomized in the experimental group will wear a virtual reality headset diffusing an atmosphere considered as relaxing. The expected results of this work would be a significant decrease in pain during oocyte retrieval under local anesthesia in patients wearing the virtual reality headset, associated with a decrease of anxiety and a significantly higher satisfaction score. The final objective would be to consider this tool as a non-invasive means that could be used in routine in the department of Medically Assisted Reproduction of Rennes, but also in other cities. In the longer term, the reduction of pain and anxiety could encourage patients to choose local anesthesia and therefore increase its use.

Observational, prospective, randomized, open-label, monocentric study.

ELIGIBILITY:
Inclusion Criteria:

* Female adult (at least 18 years old)
* For whom an oocyte retrieval is planned
* Who has had an anesthesia consultation
* Who has chosen local anesthesia
* Who has signed an informed and written consent
* Affiliated to a social security system.

Exclusion Criteria:

* Pre-existing dizzying sensations
* Severe facial wounds
* History of epilepsy
* Adults under legal protection, curatorship or guardianship, adults deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Reproductive Cell Retrieval
Enrollment: 90 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain during oocyte retrieval | 30 minutes
  The assessment criteria used is the numerical pain scale from 0 to 10 (0 = no pain, 10 = extremely painful)

SECONDARY OUTCOMES:
Anxiety during oocyte retrieval | 30 minutes
  The assessment criteria used a numerical scale ranging from 0 to 10 (0 = no anxiety, 10 = extremely anxious).
Immediate postoperative pain | 30 minutes
  The assessment criteria used is the numerical pain scale from 0 to 10 (0 = no pain, 10 = extremely painful)
The pain felt by the patient during the oocyte retrieval, according to the gynecologist who did the retrieval | 30 minutes
  The assessment criteria used is the numerical pain scale from 0 to 10 (0 = no pain, 10 = extremely painful)
immediate postoperative satisfaction | 30 minutes
  The assessment criteria used is the Likert scale ranging from 1 (Very dissatisfied) to 5 (Very satisfied)
Use of a complementary sedation or a general anesthesia | 30 minutes
  This criteria will be filled in by the gynecologistby the gynecologist who performed the retrieval:
  * Only local anesthesia
  * Use of an additional sedation
  * Switch to general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France